CLINICAL TRIAL: NCT02798692
Title: Randomized, Placebo-controlled, Double-blind Phase I Dose-escalating Trial to Evaluate the Safety and Immunogenicity of a Vaccine Against Human Cytomegalovirus
Brief Title: Trial to Evaluate Safety and Immunogenicity of a Vaccine Against HCMV
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Hookipa Biotech GmbH (Industry)
Collaborators: Centre for Vaccinology Ghent - CEVAC (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: H-100-001
Record Dates: First submitted 2016-06-09; First posted 2016-06-14 (Estimated); Last update posted 2018-04-03 (Actual); Status verified 2018-03

CONDITIONS: Cytomegalovirus Infection
Keywords: Prevention
MeSH Terms: conditions — Cytomegalovirus Infections

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Low dose HB-101 group (Active Comparator): Intervention:Three administrations of a low dose of HB-101
  Interventions: Biological: Low dose HB-101
- Medium dose HB-101 group (Active Comparator): Intervention:Three administrations of a middle dose of HB-101.
  Interventions: Biological: Medium dose HB-101
- High dose HB101 group (Active Comparator): Intervention:Three administrations of a high dose of HB-101.
  Interventions: Biological: High dose HB-101
- Placebo group (Placebo Comparator): Intervention:Three administrations of placebo (diluent)
  Interventions: Biological: Placebo

INTERVENTIONS:
Biological: Low dose HB-101 — Three intra muscular administrations at Day 0, Month 1 and Month 3
  Arms: Low dose HB-101 group
Biological: Medium dose HB-101 — Three intra muscular administrations at Day 0, Month 1 and Month 3
  Arms: Medium dose HB-101 group
Biological: High dose HB-101 — Three intra muscular administrations at Day 0, Month 1 and Month 3
  Arms: High dose HB101 group
Biological: Placebo — Three intra muscular administrations at Day 0, Month 1 and Month 3. The diluent is used as placebo.
  Arms: Placebo group

SUMMARY:
The objectives of this first-in-human is to evaluate the safety and the immunogenicity of three administrations of a bivalent vaccine candidate against human cytomegalovirus, at three different dose levels.

DETAILED DESCRIPTION:
Hookipa Biotech AG is developing a replication-deficient lymphocytic choriomeningitis virus (rLCMV) vector platform. HB-101 is a bivalent vaccine containing two recombinant, replication-deficient lymphocytic choriomeningitis virus (rLCMV) vectors, one expressing the pp65 protein of the human cytomegalovirus (HCMV) and one expressing the gB protein of human cytomegalovirus (HCMV).

This Phase 1 will enroll three successive cohorts of 18 healthy volunteers. Each cohort will receive either a low dose, a middle dose or a high dose of the vaccine (n=14 volunteers), or placebo (n=4). A DSMB will review the safety data for the low dose cohort, before progressing to the middle, and so before high dose. Eight DSMB meetings have been planned for the whole study.

The subjects will be followed up to 12 months post first administration.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent
* Male or female, aged 18-45 years, in good health.
* Negative for HCMV
* Body mass index between 19 and 32 kg/m²
* Willing to forego receipt of other routine vaccinations (with the exception of seasonal influenza vaccination) for five months after study entry.
* For female volunteers: use of effective birth control for at least 2 months prior to study entry and willing to use effective birth control measures up to the Month 12 visit
* Comply with the requirements of this protocol (e.g. return for follow-up visits), as judged by the Investigator.

Exclusion Criteria:

* Works as a childcare provider.
* Pregnant or breastfeeding woman.
* Any screening safety laboratory value that is 2 times above the upper limit of normal value.
* Any confirmed or suspected immunodeficiency or autoimmune disorder.
* Treatment with any chronic immunosuppressive medication or other immuno-modifying drugs within 6 months prior to study entry. However, inhaled and topical steroids are allowed.
* Any vaccination other than for seasonal influenza within 3 months prior to study entry.
* Previous vaccination with an investigational HCMV vaccine.
* Receipt of blood, blood products and/or immunoglobulins within 3 months prior to study entry.
* History of severe allergic reactions and /or anaphylaxis
* Allergy to any component of the vaccine preparation.
* Expected to be unavailable to complete study follow up.
* Tested positive for HIV, HBsAg and/or anti-HCV.
* Participating in another clinical trial.
* Subject with a rash, dermatological condition or tattoos in the area of the injection site, as these may interfere with administration site reaction rating.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 54 (Actual)
Dates: Start 2016-06 (Actual); Primary Completion 2017-05 (Actual); Study Completion 2018-03 (Actual)

PRIMARY OUTCOMES:
Safety primary outcome (local solicited symptoms) | Day 0 to Day 7 after each administration
  Local solicited symptoms will be assessed by diary card and scripted questions for 7 days after each administration: administration site pain, induration, erythema, pruritus and swelling
Safety primary outcome (general solicited symptoms) | Day 0 to Day 7 after each administration
  General solicited symptoms will be assessed by diary card and scripted questions for 7 days after each administration: malaise, fatigue, body temperature (measured axillary), generalized myalgia.
Safety primary outcome (Unsolicited AE´s) | From Day 0 to Month 4
  Unsolicited AEs will be recorded through open-ended general inquiries
Safety primary outcome (SAEs and pregnancies) | From Day 0 to Month 12
  SAEs and pregnancies will be recorded during the whole study
Safety primary outcome (Vital signs) | From Day 0 to Month 12
  Vital signs (blood pressure, heart rate and body temperature)
Safety primary outcome (physical examination) | From Day 0 to Month 12
  general evaluation based on the Investigator judgment and local evaluation of the administration site
Safety primary outcome (Clinical evaluation - part I) | From Day 0 to Month 12
  Complete blood count
Safety primary outcome (Clinical evaluation - part II) | From Day 0 to Month 12
  Comprehensive Metabolic Panel

SECONDARY OUTCOMES:
Humoral Immunogenicity | From Day 0 to Month 12
  * Human cytomegalovirus (HCMV) gB immunoglobulin G (IgG) by enzyme-linked immunosorbent assay (ELISA)
  * HCMV neutralization on MRC-5 cells
  * HCMV neutralization on ARPE-19 cells (depending on neutralization assay results in MRC-5 cells)
  * Lymphocytic choriomeningitis virus (LCMV) neutralization on ARPE-19 cells
Cellular Immunogenicity | From Day 0 to Month 12
  * LCMV NP-specific interferon γ (IFN-γ) Enzyme-Linked Immunospot Assay (ELISPOT)
  * LCMV NP-specific intracellular cytokine staining (ICS) of CD4+ and CD8+ T cells for IFN-γ, IL-2, TNF-α, CD107a and CD40L
  * HCMV pp65-specific IFN-γ ELISPOT
  * HCMV gB-specific IFN-γ ELISPOT
  * HCMV pp65-specific ICS of CD4+ and CD8+ T cells for IFN-γ, IL-2, TNF-α, CD107a and CD40L
  * HCMV gB-specific ICS of CD4+ and CD8+ T cells for IFN-γ, IL-2, TNF-α, CD107a and CD40L

CONTACTS AND LOCATIONS:
Overall Officials: Geert Leroux-Roels, MD PhD Prof, Principal Investigator — UZ Gent
Locations (1):
- Center for Vaccinology Ghent, Ghent, East Flanders, Belgium

IPD SHARING:
Plan to Share IPD: No